CLINICAL TRIAL: NCT03107845
Title: Randomized Controlled Trial to Evaluate the Effects of Psychometric Feedback on Treatment Outcome and Its Mediators and Moderators in Outpatient Psychotherapy
Brief Title: Randomized Controlled Trial to Evaluate Personalized Prediction and Adaptation Tools in Psychotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trier (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Prof. Dr. Wolfgang Lutz, Prof. Dr. Wolfgang Lutz, University of Trier
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LU 660/10-1
Record Dates: First submitted 2017-03-30; First posted 2017-04-11 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Feedback, Psychological
Keywords: CBT; Psychometric Feedback; Clinical Support Tools; Personalized Mental Health
MeSH Terms: interventions — Cognitive Behavioral Therapy; galactosylceramide sulfotransferase

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cognitive Behavior Therapy (Active Comparator): Cognitive Behavioral Therapy without psychometric Feedback.
  Interventions: Behavioral: Cognitive Behavior Therapy
- CBT plus Feedback (Experimental): Cognitive Behavioral Therapy (CBT) with Psychometric Feedback
  Interventions: Behavioral: CBT plus Feedback
- CBT plus Feedback plus CST (Experimental): Cognitive Behavioral Therapy (CBT) with Psychometric Feedback and Clinical Support Tools (CST)
  Interventions: Behavioral: CBT plus Feedback plus CST

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy — Treatments are conducted by cognitive-behavioral therapists in training with different levels of experience as well as licensed cognitive-behavioral therapists with several years of experience. The treatment approach is based on cognitive-behavioral manuals and principles.
  Arms: Cognitive Behavior Therapy
Behavioral: CBT plus Feedback — Therapists of the IG1 are provided with information about the initial status concerning symptoms (BSI & OQ-30), interpersonal functioning (IIP-32 & OQ-30) as well as diagnoses specific symptoms (GAD-7 or PHQ-9). Beside the status measures, also individual progress information on the symptom level (HSCL-11 each session) is provided to the therapist. Randomized controlled trial to evaluate the effects of personalized prediction and adaptation tools on treatment outcome in outpatient psychotherapy. This group is a matched sample.
  Arms: CBT plus Feedback
Behavioral: CBT plus Feedback plus CST — Additional to the intervention group "CBT and Feedback" therapists will be provided with additional clinical support tools (CST) which are designed to facilitate treatment selection and treatment adaptation. The causes of deterioration will be assessed and therapists will be provided with additional treatment recommendations and material to help preventing treatment failure for a specific patient. During treatment the clinical support tools will be provided in the problem fields: risk/suicidality, motivation / treatment goals, therapeutic relationship, social support / critical life events, and emotion regulation / self regulation.
  Arms: CBT plus Feedback plus CST

SUMMARY:
The research project investigates in a randomized controlled trial the effectiveness as well as moderating and mediating factors of psychometric feedback to therapists. In the intended study a total of 423 patients, who applied for a cognitive-behavioral therapy at the psychotherapy clinic of the University Trier and suffer from a depressive and/or an anxiety disorder (SCID-interviews), will be included. The patients will be randomly assigned either to one therapist as well as to one of two intervention groups (CG, IG2). An additional intervention group (IG1) will be generated from an existing archivale data set via propensity score matching. Patients of the control group (CG; n = 85) will be monitored concerning psychological impairment but therapists will not be provided with any feedback about the patients assessments. In both intervention groups (IG1: n = 169; IG2: n = 169) the therapists are provided with feedback about the patients self-evaluation in a computerized feedback portal. Therapists of the IG2 will additionally be provided with clinical support tools, which will be developed in this project, on the basis of existing systems. Therapists will also be provided with a personalized treatment recommendation based on similar patients (Nearest Neighbors) at the beginning of treatment.

Besides the general effectiveness of feedback and the clinical support tools for negatively developing patients, further mediating and moderating variables on this feedback effect should be examined: treatment length, frequency of feedback use, therapist effects, therapist's experience, attitude towards feedback as well as congruence of therapist's and patient's evaluation concerning the progress.

Additional procedures will be implemented to assess treatment adherence as well as the reliability of diagnosis and to include it into the analyses.

DETAILED DESCRIPTION:
The primary objective of the current project is to investigate several questions of feedback research in psychotherapy with a cluster randomized controlled trial (RCT) with two feedback groups (IG1: Feedback; IG2: Feedback plus CSTs) and one CG with repeated measurements. IG1 will be generated from an existing archival data set via propensity score matching. It adds to previous feedback research a stricter design by investigating another repeated measurement CG as well as a stricter control of treatment integrity. It also includes a structured clinical interview (SCID) and controls for comorbidity (within depression and anxiety). Furthermore, a more severely impaired patient sample is studied and an international outcome instrument is used, which is also often applied in outpatient centers in Germany. This study also investigates the above described moderators (attitudes towards, use of the feedback system, diagnoses) and mediators (therapists' awareness of negative change and treatment length) in a comprehensive model and in one study.

Therefore, the research questions are:

Main questions:

H1: NOT patients in the feedback condition (IG1) show on average better treatment outcome than NOT patients in the CG.

H2: NOT patients in the IG2 (+CSTs) show on average better treatment outcomes than NOT patients of the IG1 (no CSTs but psychometric feedback).

Secondary questions concerning moderators and mediators:

H3: The positive impact of feedback for NOT patients is moderated through the usage of the feedback system and/or the attitudes of the therapist towards feedback.

* H3a: The more frequently and the longer feedback is used, the more aware are therapists for negative change.
* H3b: The more positive the therapists' attitudes towards, the more aware are therapists for negative change.
* H3c: The effects of feedback on patient outcomes do not differ between diagnostic groups (depression and anxiety).

H4: The positive impact of feedback for NOT patients is mediated through therapists' awareness of negative change as well as treatment length

* H4a: The positive impact of feedback for NOT patients is mediated by the therapists' awareness of negative developments of patients.
* H4b: The positive effect of therapists' awareness on treatment outcome is mediated by treatment length (number of sessions).

It is assumed that feedback raises therapists' awareness of negative change. This increased awareness could directly improve treatment outcome through a respective treatment adaption. Given the finding that NOT patients tend to have longer treatments when therapists receive feedback, this effect of increased awareness on treatment outcome could be mediated through treatment length. Accordingly, the essential adaption after being aware of a negative progress would be a higher number of sessions which gives NOT patients more time to improve. However, other adaptions than an increased treatment length are possible and could directly enhance treatment outcome. Regarding the above described moderators it is assumed that the amount of feedback induced awareness as well as the positive effect of feedback on outcome is potentially influenced by therapists' attitude towards feedback, the usage of the feedback system and diagnoses.

Furthermore, effects of feedback are controlled for the following potential influence factors: treatment integrity (adherence, competence), comorbidity, initial impairment, clinical experience as well as experience with the feedback system, non-psychometric feedback and therapist effects (Level 2 variable).

To answer these questions, the following treatment and CSTs will be studied in the outpatient clinic at the University of Trier:

* Control group (CG): Treatment with continuous assessments but without computer based feedback to therapists.
* Intervention group 1(IG1): Treatment with continuous assessments including computer based feedback to therapists after each session. This group is a matched sample.
* Intervention group 2(IG2): Treatment with continuous assessments including computer based feedback to therapists after each session including an alarm for NOT patients and the provision of CST for NOT patients.

ELIGIBILITY:
Inclusion Criteria:

* One anxiety and/or depressive disorder (ICD-10: F32, F33, F40, F41, F42, F43)
* At least 3 treatment sessions

Exclusion Criteria:

* Organic, including symptomatic mental disorders (ICD-10: F00-F09)
* Mental and behavioral disorders due to psychoactive substances (ICD-10: F10-F19)
* Schizophrenia, schizotypal, and delusional disorders (ICD-10: F20-F29)
* Acute suicidality

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 423 (Actual)
Dates: Start 2017-04-15 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Change in 11-item Short version of Hopkins' Symptom Checklist (HSCL-11; Lutz, Tholen, Schürch, & Berking, 2006) | through study completion, an average of 50 weeks
  The mean of the HSCL-11 is used as the main outcome measure administered before each session.

SECONDARY OUTCOMES:
Change in Outcome Questionnaire (OQ-30; Lambert et al., 1996) | through study completion, an average of 50 weeks
  The mean of the OQ-30 is used as the secondary outcome measure administered every fifth session.
Change in Patient Health Questionnaire (PHQ-9; Kroenke, Spitzer, & Williams, 2001) | through study completion, an average of 50 weeks
  The sum of the PHQ-9 is used as the secondary outcome measure administered every fifth session.
Change in Generalized Anxiety Disorder (GAD-7; Spitzer, Kroenke, Williams, & Löwe, 2006) | through study completion, an average of 50 weeks
  The sum of the GAD-7 is used as the secondary outcome measure administered every fifth session.
Change in the Brief Symptom Inventory (BSI; Franke, 2000) | through study completion, an average of 50 weeks
  The GSI of the BSI is used as a secondary outcome measure administered at the beginning and the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Lutz, Prof. Dr., Principal Investigator — University of Trier
Locations (1):
- University of Trier, Trier, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lutz W, De Jong K, Rubel J. Patient-focused and feedback research in psychotherapy: Where are we and where do we want to go? Psychother Res. 2015;25(6):625-32. doi: 10.1080/10503307.2015.1079661. Epub 2015 Sep 16. PMID 26376225
- [Background] Lutz W, Rubel J, Schiefele AK, Zimmermann D, Bohnke JR, Wittmann WW. Feedback and therapist effects in the context of treatment outcome and treatment length. Psychother Res. 2015;25(6):647-60. doi: 10.1080/10503307.2015.1053553. Epub 2015 Jul 28. PMID 26218788
- [Derived] Lutz W, Zimmermann D, Muller VNLS, Deisenhofer AK, Rubel JA. Randomized controlled trial to evaluate the effects of personalized prediction and adaptation tools on treatment outcome in outpatient psychotherapy: study protocol. BMC Psychiatry. 2017 Aug 24;17(1):306. doi: 10.1186/s12888-017-1464-2. PMID 28836954